CLINICAL TRIAL: NCT03072576
Title: A Multicentre Study of the Diagnostic Accuracy and Feasibility of the Xpert Ultra for Detection of TB and Rifampin Resistance in Adults Suspected of Having Pulmonary TB
Brief Title: Accuracy and Feasibility of Xpert Ultra
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 7210-04-2/1
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Diagnosis; Xpert MTB/RIF; Ultra Xpert MTB/RIF
MeSH Terms: conditions — Tuberculosis, Pulmonary; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Xpert MTB/RIF Ultra — Next generation Xpert MTB/RIF assay, this cartridge is intended for the detection of M. tuberculosis in sputum as well as the detection of M. tuberculosis mutations associated with resistance to rifampin
  Other Names: Cepheid Ultra

SUMMARY:
Consenting adults presenting with signs and symptoms compatible with pulmonary tuberculosis will be interviewed for demographic and medical information, and then will be asked to provide 3-4 expectorated sputum specimens. In the study laboratory, sputa will be tested using conventional and investigational diagnostic tests for tuberculosis and rifampin resistance.

ELIGIBILITY:
Case Detection Group

Inclusion Criteria:

* Age 18 years or above;
* Provision of informed consent;
* Willingness to provide 4 sputum specimens at enrolment;
* Willingness to have a study follow-up visit approximately 42 to 70 days after enrolment
* Clinical suspicion of pulmonary TB (including cough ≥2 weeks and at least 1 other symptom typical of TB)

Exclusion Criteria:

* Receipt of any dose of TB treatment within 6 months prior to enrolment
* Participants for whom, at the time of enrolment, the follow-up visit is judged to be poorly feasible (e.g. individuals planning to relocate)

Drug-Resistant TB Group

Inclusion Criteria:

* Age 18 years or above;
* Provision of informed consent;
* Willingness to provide 4 sputum specimens at enrolment;
* Non-converting pulmonary TB cases (category I and category II failures) or multi-drug resistant (MDR) suspect* (based on World Health Organization definition), i.e. at least one of the following: i) retreatment cases, ii) active TB cases that are MDR-contacts and iii) patients at high risk for MDR-TB as determined by local program (e.g. prisoners)

Exclusion Criteria:

• none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have symptoms consistent with pulmonary TB presenting to participating centres.
  Two groups of participants will be recruited, namely a 'Case Detection Group' and a 'Drug-Resistant TB Group'.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Difference in sensitivity and specificity (ability to correctly identify those with TB and those without TB) between Xpert Ultra and Xpert MTB/ for Mycobacterium tuberculosis (MTB) detection (non-inferiority endpoint) | Day 1

SECONDARY OUTCOMES:
Sensitivity of Xpert Ultra for MTB detection (ability to correctly identify those with TB i.e. true positives), stratified by smear status | Day 1
Sensitivity and specificity (ability to correctly identify those with TB resistant to Rifampin and those with TB susceptible to Rifampin) of Xpert Ultra for detection of Rifampin (RIF) resistance | Day 1
Difference in sensitivity and specificity (ability to correctly identify those with TB resistant to Rifampin and those with TB susceptible to Rifampin) of Xpert Ultra and Xpert MTB/RIF for detection of RIF resistance | Day 1
Proportion of test attempts that do not yield a determinate result for Xpert Ultra and for Xpert MTB/RIF | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Denkinger, MD, PhD, Principal Investigator — Find
Locations (6):
- Republican Research and Practical Centre for Pulmonology and Tuberculosis, Minsk, Belarus
- Clinical Research Unit, National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- India (3):
  - National Institute for Research in Tuberculosis, Madras
  - Dept of Microbiology, Hinduja Hospital, Mumbai
  - New Delhi Tuberculosis Centre, New Delhi
- Department of Molecular Medicine and Haematology, School of Pathology, Faculty of Health Science, University of the Witwatersrand, and The National Priority Program of the National Health Laboratory Service, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Undecided